# Phase II Study of Pembrolizumab and Lenvatinib in Advanced Well-Differentiated Neuroendocrine Tumors

NCT03290079

Version 5.0

December 10, 2018



**SPONSOR:** Merck

TITLE: Phase II study of pembrolizumab and lenvatinib in advanced well-differentiated neuroendocrine tumors

**IND NUMBER: 135156** 

# **Principal Investigator**

Jonathan Strosberg, MD H. Lee Moffitt Cancer Center, 12902 Magnolia Dr. Tampa, FL 33612 jonathan.strosberg@moffitt.org

Phone: 813-745-3636 Fax: 813-745-7229

# Statistician:

1

Michael Schell, PhD H. Lee Moffitt Cancer Center, 12902 Magnolia Dr. Tampa, FL 33612 michael.schell@moffitt.org

Phone: 813-745-6061 Fax: 813-745-5855



# **Table of contents**

| Tl | RIAL DESIGN | 5 |
|---|---|---|
| O | BJECTIVES & HYPOTHESES | 5 |
| .1 | Primary Objective & Hypothesis | 5 |
| .2 | Secondary Objectives | 5 |
| .3 | Exploratory Objective | 6 |
| BA | ACKGROUND & RATIONALE | 6 |
| .1 | Background | 6 |
| 4.1.1 | Pharmaceutical and Therapeutic Background | 6 |
| 4.1.2 | Preclinical and Clinical Trial Data | 7 |
| .2 | Rationale | 8 |
| 4.2.1 | Rationale for the Trial and Selected Subject Population | 8 |
| 4.2.2 | Rationale for Dose Selection/Regimen/Modification | 8 |
| 4.2.3 | Rationale for Endpoints | . 10 |
| M | ETHODOLOGY | . 11 |
| .1 | Entry Criteria | . 11 |
| 5.1.1 | Diagnosis/Condition for Entry into the Trial | . 11 |
| 5.1.2 | Subject Inclusion Criteria | . 11 |
| 5.1.3 | Subject Exclusion Criteria | . 13 |
| .2 | Trial Treatments | . 15 |
| 5.2.1 | Dose Selection/Modification | . 16 |
| 5.2.2 | Timing of Dose Administration | . 24 |
| 5.2.3 | Trial Blinding/Masking | . 25 |
| | Ol. 1.1 2.2 3.3 BA 4.1.1 4.1.2 2.4.2.1 4.2.2 4.2.3 M 5.1.1 5.1.2 5.1.3 2.5 5.2.2 | 2 Secondary Objectives BACKGROUND & RATIONALE |



| 5. | .3 | Concomitant Medications/Vaccinations (allowed & prohibited) | . 25 |
|---|---|---|---|
| | 5.3.1 | Acceptable Concomitant Medications | . 25 |
| | 5.3.2 | Prohibited Concomitant Medications | . 25 |
| 5. | .4 | Diet/Activity/Other Considerations | . 26 |
| | 5.4.1 | Diet | . 26 |
| | 5.4.2 | Contraception | . 26 |
| | 5.4.3 | Use in Pregnancy | . 28 |
| | 5.4.4 | Use in Nursing Women | . 29 |
| 5. | .5 | Subject Withdrawal/Discontinuation Criteria | . 29 |
| 5. | .6 | Subject Replacement Strategy | . 30 |
| 5. | .7 | Clinical Criteria for Early Trial Termination | . 30 |
| 6.0 | TF | RIAL FLOW CHART | . 31 |
| 6. | .1 | Study Flow Chart | . 31 |
| 7.0 | TF | RIAL PROCEDURES | . 33 |
| 7. | .1 | Trial Procedures | . 33 |
| | 7.1.1 | Administrative Procedures | . 33 |
| | 7.1.2 | Clinical Procedures/Assessments | . 35 |
| | 7.1.3 | Laboratory Procedures/Assessments | . 36 |
| | 7.1.4 | Other Procedures | . 38 |
| | 7.1.5 | Visit Requirements | . 38 |
| 7. | .2 | Assessing and Recording Adverse Events | . 39 |
| | 7.2.1 | Definition of an Overdose for This Protocol and Reporting of Overdose to the Sponsor and to Merck | . 40 |



| | 7.2 | 2.2 | Reporting of Pregnancy and Lactation to the Sponsor and to Merck | 41 |
|---|---|---|---|---|
| | 7.2 | 2.3 | Immediate Reporting of Adverse Events to the Sponsor and to Merck | 41 |
| | 7.2 | 2.4 | Evaluating Adverse Events | 44 |
| | 7.2 | 2.5 | Sponsor Responsibility for Reporting Adverse Events | 48 |
| 8.0 | , | STA | ATISTICAL ANALYSIS PLAN | 48 |
| 8 | 8.1 | S | tatistical Analysis Plan Summary | 48 |
| 8 | 8.2 | S | tatistical Analysis Plan | 48 |
| 9.0 | | | BELING, PACKAGING, STORAGE AND RETURN OF CLINICAL PPLIES | . 48 |
| 9 | 9.1 | Iı | nvestigational Product | 48 |
| 9 | 9.2 | P | Packaging and Labeling Information | 49 |
| 9 | 9.3 | C | Clinical Supplies Disclosure | 49 |
| 9 | 9.4 | S | torage and Handling Requirements | 49 |
| 9 | 9.5 | R | Returns and Reconciliation | 49 |
| 10. | .0 | AD | MINISTRATIVE AND REGULATORY DETAILS | . 50 |
| | 10.1 | C | Compliance with Trial Registration and Results Posting Requirements | 50 |
| | 10.2 | D | Oata Management | 50 |
| 11. | .0 | API | PENDICES | 51 |
| | 11.1 | E | CCOG Performance Status | 51 |
| | 11.2 | C | Common Terminology Criteria for Adverse Events V4.0 (CTCAE) | 51 |
| | 11.3 | | Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 Criteria for Evaluating Response in Solid Tumors | . 51 |
| 12. | .0 | REI | FERENCES | . 52 |



### 1.0 TRIAL SUMMARY

| Abbreviated Title | Pembrolizumab in advanced well-differentiated neuroendocrine tumors |
|---|---|
| Trial Phase | II |
| Clinical Indication | Metastatic progressive neuroendocrine tumors of lung, thymic, small bowel, colorectal and unknown primary origin |
| Trial Type | Single arm, phase II Simon 2-stage design |
| Type of control | N/A |
| Route of administration | IV |
| Trial Blinding | N/A |
| Treatment Groups | N/A |
| Number of trial subjects | 35 |
| Estimated enrollment period | 24 months |
| Estimated duration of trial | 4 years |
| Duration of Participation | 2 years |
| Estimated average length of treatment per patient | 9 months |

### 2.0 TRIAL DESIGN

Trial Design: 2-stage, single arm, open-label phase II study

### 3.0 OBJECTIVES & HYPOTHESES

# 3.1 Primary Objective & Hypothesis

• **Objective**: To assess the overall radiographic response rate (ORR) associated with pembrolizumab in patients with advanced, progressive well-differentiated neuroendocrine tumors

**Hypothesis:** Well-differentiated neuroendocrine tumors (any grade) will be sensitive to combination VEGF and PD-1 inhibition resulting in a clinically meaningful response rate

# 3.2 Secondary Objectives

- **Objective**: To assess progression-free survival (PFS) in this population based on RECIST 1.1
- **Objective**: To assess duration of response (DOR) by RECIST 1.1
- Objective: To assess overall survival (OS) in this population
- Objective: To assess safety and tolerability



# 3.3 Exploratory Objective

• **Objective:** Correlate response with PD-L1 tumor expression, tumor mutation burden (TMB), and MSI status

### 4.0 BACKGROUND & RATIONALE

# 4.1 Background

Refer to the Investigator's Brochures (IB)/approved labeling for detailed background information on pembrolizumab and lenvatinib.

# 4.1.1 Pharmaceutical and Therapeutic Background

#### 4.1.1.1 Pembrolizumab

The importance of intact immune surveillance in controlling outgrowth of neoplastic transformation has been known for decades. Accumulating evidence shows a correlation between tumor-infiltrating lymphocytes (TILs) in cancer tissue and favorable prognosis in various malignancies. In particular, the presence of CD8+ T-cells and the ratio of CD8+ effector T-cells / FoxP3+ regulatory T-cells seems to correlate with improved prognosis and long-term survival in many solid tumors.

The PD-1 receptor-ligand interaction is a major pathway hijacked by tumors to suppress immune control. The normal function of PD-1, expressed on the cell surface of activated Tcells under healthy conditions, is to down-modulate unwanted or excessive immune responses, including autoimmune reactions. PD-1 (encoded by the gene Pdcd1) is an Ig superfamily member related to CD28 and CTLA-4 which has been shown to negatively regulate antigen receptor signaling upon engagement of its ligands (PD-L1 and/or PD-L2). The structure of murine PD-1 has been resolved. PD-1 and family members are type I transmembrane glycoproteins containing an Ig Variable-type (V-type) domain responsible for ligand binding and a cytoplasmic tail which is responsible for the binding of signaling molecules. The cytoplasmic tail of PD-1 contains 2 tyrosine-based signaling motifs, an immunoreceptor tyrosine-based inhibition motif (ITIM) and an immunoreceptor tyrosine-Following T-cell stimulation, PD-1 recruits the tyrosine based switch motif (ITSM). phosphatases SHP-1 and SHP-2 to the ITSM motif within its cytoplasmic tail, leading to the dephosphorylation of effector molecules such as CD3ζ, PKCθ and ZAP70 which are involved in the CD3 T-cell signaling cascade. The mechanism by which PD-1 down modulates T-cell responses is similar to, but distinct from that of CTLA-4 as both molecules



regulate an overlapping set of signaling proteins. PD-1 was shown to be expressed on activated lymphocytes including peripheral CD4+ and CD8+ T-cells, B-cells, T regs and Natural Killer cells. Expression has also been shown during thymic development on CD4-CD8- (double negative) T-cells as well as subsets of macrophages and dendritic cells. The ligands for PD-1 (PD-L1 and PD-L2) are constitutively expressed or can be induced in a variety of cell types, including non-hematopoietic tissues as well as in various tumors. Both ligands are type I transmembrane receptors containing both IgV- and IgC-like domains in the extracellular region and contain short cytoplasmic regions with no known signaling motifs. Binding of either PD-1 ligand to PD-1 inhibits T-cell activation triggered through the T-cell receptor. PD-L1 is expressed at low levels on various non-hematopoietic tissues, most notably on vascular endothelium, whereas PD-L2 protein is only detectably expressed on antigen-presenting cells found in lymphoid tissue or chronic inflammatory environments. PD-L2 is thought to control immune T-cell activation in lymphoid organs, whereas PD-L1 serves to dampen unwarranted T-cell function in peripheral tissues. Although healthy organs express little (if any) PD-L1, a variety of cancers were demonstrated to express abundant levels of this T-cell inhibitor. PD-1 has been suggested to regulate tumor-specific T-cell expansion in subjects with melanoma (MEL). This suggests that the PD-1/PD-L1 pathway plays a critical role in tumor immune evasion and should be considered as an attractive target for therapeutic intervention.

Pembrolizumab is a potent and highly selective humanized monoclonal antibody (mAb) of the IgG4/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2. Keytruda® (pembrolizumab) has been approved in the United States for the treatment of patients non-small cell lung cancer (1<sup>st</sup> and 2<sup>nd</sup> line), head and neck cancer, and melanoma.

#### 4.1.1.2 Lenvatinib

Lenvatinib is a receptor tyrosine kinase (RTK) inhibitor that inhibits the kinase activities of vascular endothelial growth factor (VEGF) receptors VEGFR1 (FLT1), VEGFR2 (KDR), and VEGFR3 (FLT4). Lenvatinib also inhibits other RTKs that have been implicated in pathogenic angiogenesis, tumor growth, and cancer progression in addition to their normal cellular functions, including fibroblast growth factor (FGF) receptors FGFR1, 2, 3, and 4; the platelet derived growth factor receptor alpha (PDGFRα), KIT, and RET.

# 4.1.2 Preclinical and Clinical Trial Data

Refer to the Investigator's Brochures and package inserts for Preclinical and Clinical data.



#### 4.2 Rationale

# 4.2.1 Rationale for the Trial and Selected Subject Population

The treatment landscape of advanced neuroendocrine tumors (NET) has advanced rapidly in the past decade, with several systemic therapeutic options for patients with metastatic disease. However, immunotherapy drugs have not been shown to be highly active in well-differentiated gastroenteropancreatic or lung NETs, or in poorly differentiated neuroendocrine carcinomas originating outside the lung. Preliminary evidence suggests that PD-1 inhibitor monotherapy is relatively ineffective, with response rates <10% in most subsets of NETs.

Lenvatinib, a multitargeted tyrosine kinase inhibitor (TKI) which inhibits the kinase activities of vascular endothelial growth factor (VEGF) receptors VEGFR1 (FLT1), VEGFR2 (KDR), and VEGFR3 (FLT4) has been recently reported to be effective in NETs progressing after several lines of therapy (ESMO). Response rates were 40% in pancreatic NETs, and 18.5% in gastrointestinal NETs.<sup>8</sup>

Recent data supports the hypothesis that combining antiangiogenic treatment with immune checkpoint inhibition can be synergistic. Several trials have been conducted evaluating the combinations of antiangiogenic agents with checkpoint inhibitors in renal cell carcinoma (mRCC) and anaplastic thyroid carcinoma (ATC) with promising results<sup>9-12</sup>. Checkmate-016, comparing nivolumab + sunitinib and nivolumab + pazopanib showed an ORR of 52 and 45%, and a PFS of 48.9 and 31.4 months, respectively. A study evaluating pembrolizumab and lenvatinib in mRCC showed an ORR of 69%, with half of the patients exhibiting PR. Lenvatinib plus pembrolizumab has shown striking results in endometrial cancer. In a phase Ib/II basket study (KEYNOTE 146 trial; NCT02501096), of heavily pretreated patients, ORR at week 24 was 45% and the overall ORR was 47.2%. This study led the FDA to grant a breakthrough therapy designation for the combination of lenvatinib and pembrolizumab in 8/2018.

Given the encouraging results in other trials, and the fact that VEGFR-TKIs typically produce fast but non-durable responses and checkpoint inhibitors produce slow but durable responses, this is combination therapy is of particular interest to explore in NET tumors. Pancreatic NETs will be excluded due to the already high response rate observed with lenvatinib monotherapy.

# 4.2.2 Rationale for Dose Selection/Regimen/Modification

# 4.2.2.1 Pembrolizumab

An open-label Phase I trial (Protocol 001) was conducted to evaluate the safety and clinical activity of single agent pembrolizumab. The dose escalation portion of this trial evaluated three dose levels, 1 mg/kg, 3 mg/kg, and 10 mg/kg, administered every 2 weeks (Q2W) in



subjects with advanced solid tumors. All three dose levels were well tolerated and no dose-limiting toxicities were observed. This first in human study of pembrolizumab showed evidence of target engagement and objective evidence of tumor size reduction at all dose levels (1 mg/kg, 3 mg/kg and 10 mg/kg Q2W). No MTD has been identified to date. 10.0 mg/kg Q2W, the highest dose tested in PN001, will be the dose and schedule utilized in Cohorts A, B, C and D of this protocol to test for initial tumor activity. Recent data from other clinical studies within the pembrolizumab program has shown that a lower dose of pembrolizumab and a less frequent schedule may be sufficient for target engagement and clinical activity.

PK data analysis of pembrolizumab administered Q2W and Q3W showed slow systemic clearance, limited volume of distribution, and a long half-life (refer to IB). Pharmacodynamic data (IL-2 release assay) suggested that peripheral target engagement is durable (>21 days). This early PK and pharmacodynamic data provides scientific rationale for testing a Q2W and Q3W dosing schedule.

A population pharmacokinetic analysis has been performed using serum concentration time data from 476 patients. Within the resulting population PK model, clearance and volume parameters of pembrolizumab were found to be dependent on body weight. The relationship between clearance and body weight, with an allometric exponent of 0.59, is within the range observed for other antibodies and would support both body weight normalized dosing or a fixed dose across all body weights. Pembrolizumab has been found to have a wide therapeutic range based on the melanoma indication. The differences in exposure for a 200 mg fixed dose regimen relative to a 2 mg/kg Q3W body weight based regimen are anticipated to remain well within the established exposure margins of 0.5 – 5.0 for pembrolizumab in the melanoma indication. The exposure margins are based on the notion of similar efficacy and safety in melanoma at 10 mg/kg Q3W vs. the proposed dose regimen of 2 mg/kg Q3W (i.e. 5-fold higher dose and exposure). The population PK evaluation revealed that there was no significant impact of tumor burden on exposure. In addition, exposure was similar between the NSCLC and melanoma indications. Therefore, there are no anticipated changes in exposure between different indication settings.

The rationale for further exploration of 2 mg/kg and comparable doses of pembrolizumab in solid tumors is based on: 1) similar efficacy and safety of pembrolizumab when dosed at either 2 mg/kg or 10 mg/kg Q3W in melanoma patients, 2) the flat exposure-response relationships of pembrolizumab for both efficacy and safety in the dose ranges of 2 mg/kg Q3W to 10 mg/kg Q3W, 3) the lack of effect of tumor burden or indication on distribution behavior of pembrolizumab (as assessed by the population PK model) and 4) the assumption that the dynamics of pembrolizumab target engagement will not vary meaningfully with tumor type.

The choice of the 200 mg Q3W as an appropriate dose for the switch to fixed dosing is based on simulations performed using the population PK model of pembrolizumab showing that the v5 dated 10Dec2018



fixed dose of 200 mg every 3 weeks will provide exposures that 1) are optimally consistent with those obtained with the 2 mg/kg dose every 3 weeks, 2) will maintain individual patient exposures in the exposure range established in melanoma as associated with maximal efficacy response and 3) will maintain individual patients exposure in the exposure range established in melanoma that are well tolerated and safe.

A fixed dose regimen will simplify the dosing regimen to be more convenient for physicians and to reduce potential for dosing errors. A fixed dosing scheme will also reduce complexity in the logistical chain at treatment facilities and reduce wastage.

#### 4.2.2.2 Lenvatinib

The recommended daily dose of lenvatinib is 24 mg (two 10mg capsules and one 4mg capsule) orally taken once daily with or without food. Lenvatinib is taken at the same time each day. If a dose is missed and cannot be taken within 12 hours, patients should skip that dose and take the next dose at the usual time of administration.

After oral administration of lenvatinib, time to peak plasma concentration (Tmax) typically occurred from 1 to 4 hours post-dose. Administration with food did not affect the extent of absorption, but decreased the rate of absorption and delayed the median Tmax from 2 hours to 4 hours.

# 4.2.3 Rationale for Endpoints

#### 4.2.3.1 Efficacy Endpoints

#### 4.2.3.1.1 Primary endpoint: RECIST-based response rate

Objective radiographic response (ORR) rate is a simple and standard criterion for assessing the efficacy of an agent(s) in a single-arm phase II trial. Numerous prior studies of pembrolizumab and lenvatinib have indicated that these agents are capable of yielding a clinically meaningful objective response in immunosensitive malignancies. Therefore ORR will be used as the primary endpoint per RECIST 1.1 criteria (see section 11.3).

# 4.2.3.1.2 Secondary efficacy endpoints

10

Secondary endpoints include: (1) DOR, defined as the time from first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first, (2) PFS, defined as the time from initial treatment to the first documented disease progression according to RECIST 1.1, or death due to any cause, whichever occurs first, and (3) OS defined as the time from initial treatment until death from any cause.

Confirmation of PR/CR should be performed with radiographic assessment  $\geq$  4 weeks after initial documentation of PR/CR.



#### 4.2.3.2 Biomarker Research

While tumoral PD-L1 expression has not been validated as a predictive marker across all malignancies, it appears to be a predictive marker for PD-1 inhibitors in some malignancies. We have previously found that well-differentiated neuroendocrine tumors can express PD-L1 (unpublished data). We will assess PD-L1 expression on archival tissue in this study both to evaluate the rate of expression of this antigen and also to analyze correlation between expression and response.

Responses to pembrolizumab have been particularly high in microsatellite instability high (MSI-H) tumors. We will therefore test for MSI status by first screening for mismatch repair (MMR) deficiency via immunohistochemical (IHC) stains. Cases that are positive for MMR protein deficiency will subsequently be tested for MSI. The prevalence of MSI-H tumors in this population of patients is unknown.

Tumor mutation burden (TMB) has emerged as a highly promising and clinically validated biomarker, particularly in the setting of lung cancer. Studies have shown that patients with high TMB can predict response to a range of various types of immunotherapy. The relationship between tumor DNA mutation burden and response to treatment will be explored.

#### 5.0 METHODOLOGY

### 5.1 Entry Criteria

### 5.1.1 Diagnosis/Condition for Entry into the Trial

Metastatic well differentiated neuroendocrine tumors of primary lung, thymic, small bowel and colorectal origin (including unknown primary)

### 5.1.2 Subject Inclusion Criteria

In order to be eligible for participation in this trial, the subject must:

- 1. Have evidence of radiographic disease progression with scan documenting progression occurring within 8 months of signing informed consent
- 2. At least two prior lines of systemic treatment. If the only prior line of treatment was adjuvant or neoadjuvant, patient must have completed treatment within 12 months. There is no limit to number of prior therapies.
- 3. Be willing and able to provide written informed consent/assent for the trial.



- 4. Be  $\geq$  18 years of age on day of signing informed consent.
- 5. Have measurable disease based on RECIST 1.1.
- 6. Have a performance status of 0 or 1 on the ECOG Performance Scale.
- 7. Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 14 days of treatment initiation.

Table 1 Adequate Organ Function Laboratory Values

| System | Laboratory Value |
|---|---|
| Hematological | |
| Absolute neutrophil count (ANC) | ≥1,500 /mcL |
| Platelets | ≥100,000 / mcL |
| Hemoglobin | ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency |
| Tiemograam | (within 7 days of assessment) |
| Renal | |
| Serum creatinine <u>OR</u> | ≤1.5 X upper limit of normal (ULN) <u>OR</u> |
| Measured or calculated <sup>a</sup> creatinine | |
| clearance | ≥60 mL/min for subject with creatinine levels > 1.5 X |
| (GFR can also be used in place of | institutional ULN |
| creatinine or CrCl) | |
| Urine protein | <30mg/dL on urinalysis or ≤1g/24 hours on 24-hour urine |
| | protein for patients with >30mg/dL on urinalysis |
| Hepatic | |
| Serum total bilirubin | ≤ 1.5 X ULN <u>OR</u> |
| | Direct bilirubin ≤ ULN for subjects with total bilirubin levels > |
| | 1.5 ULN |
| AST (SGOT) and ALT (SGPT) | ≤ 2.5 X ULN <u>OR</u> |
| AST (SGOT) and ALT (SGLT) | ≤ 5 X ULN for subjects with liver metastases |
| Albumin | ≥2.5 mg/dL |
| Coagulation | |
| International Normalized Ratio (INR) or | ≤1.5 X ULN unless subject is receiving anticoagulant therapy |
| Prothrombin Time (PT) | as long as PT or PTT is within therapeutic range of intended use |
| Frounding Time (F1) | of anticoagulants |
| Activated Partial Thromboplastin Time | ≤1.5 X ULN unless subject is receiving anticoagulant therapy |
| (aPTT) | as long as PT or PTT is within therapeutic range of intended use |
| <u> </u> | of anticoagulants |
| <sup>a</sup> Creatinine clearance should be calculated | per institutional standard. |

- 8. Female subject of childbearing potential should have a negative serum pregnancy within 72 hours prior to receiving the first dose of study medication.
- 9. Female subjects of childbearing potential (Section 5.7.2) must be willing to use an adequate method of contraception as outlined in Section 5.7.2 Contraception, for the course of the study through 120 days after the last dose of study medication.



Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

10. Male subjects of childbearing potential (Section 5.7.1) must agree to use an adequate method of contraception as outlined in Section 5.7.1- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

# 5.1.3 Subject Exclusion Criteria

The subject must be excluded from participating in the trial if the subject:

- 1. Has a poorly differentiated neuroendocrine carcinoma
- 2. Has a pancreatic neuroendocrine tumor
- 3. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
- 4. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
- 5. Has a known history of active TB (Bacillus Tuberculosis)
- 6. Hypersensitivity to pembrolizumab or any of its excipients.
- 7. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
- 8. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
  - Note: Subjects with  $\leq$  Grade 2 neuropathy are an exception to this criterion and may qualify for the study.



- Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
- 9. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
- 10. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
- 11. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
- 12. Has a history of (non-infectious) pneumonitis that required steroids, or current pneumonitis.
- 13. Has an active infection requiring systemic therapy.

14

- 14. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
- 15. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
- 16. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
- 17. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
- 18. Has received prior therapy with a tyrosine kinase inhibitor (TKI). (e.g., sunitinib, pazopanib, cabozantinib)



- 19. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
- 20. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
- 21. Has received a live vaccine within 30 days of planned start of study therapy.

Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

- 22. Uncontrolled hypertension defined as systolic blood pressure >150 mmHg or diastolic pressure >90 mmHg, despite optimal medical management.
- 23. Thrombotic or embolic events such as a cerebrovascular accident including transient ischemic, attacks, DVT within the past 6 months
- 24. Bleeding or thrombotic disorders or use of anticoagulants, such as warfarin, or similar agents requiring therapeutic international normalized ration (INR) monitoring.(Treatment with low molecular weight heparin (LMWH) is allowed)
- 25. Marked baseline prolongation of QT/QTc interval (QTc interval ≥ 500 msec) using the Fridericia method (QTc = QT/RR0.33) for QTc analysis
- 26. Clinically significant bleeding within 4 weeks
- 27. Medical need for the continued use of potent inhibitors/inducers of CYP3A4
- 28. Creatinine clearance <30 mL/min
- 29. Any condition that impairs patient's ability to swallow whole pills or gastrointestinal malabsorption that, in the investigator's opinion, might affect absorption of lenvatinib

#### 5.2 Trial Treatments

The treatment to be used in this trial is outlined below in Table 2

Table 2 Trial Treatment

| Drug | Dose/Potency | Dose | Route of | Regimen/Treatment | Use |
|---|---|---|---|---|---|
| | | Frequency | Administration | Period | |
| Pembrolizumab | 200 mg | Q3W | IV infusion | Day 1 of each 3 week cycle | Experimental |
| Lenvatinib | 24mg | QD | PO | Every day of each 3 week cycle | Experimental |

15 v5 dated 10Dec2018



Trial treatment should begin as close as possible to the date on which treatment is allocated/assigned.

### 5.2.1 Dose Selection/Modification

#### **5.2.1.1** Dose Selection

The rationale for selection of doses to be used in this trial is provided in Section 4.0 – Background and Rationale.

Details on preparation and administration of pembrolizumab and lenvatinib are provided in the Pharmacy Manuals.

# 5.2.1.2 Dose Delays and Discontinuation

Pembrolizumab and lenvatinib may be interrupted for situations other than treatment-related AEs such as medical / surgical events or logistical reasons not related to study therapy. Subjects should be placed back on study therapy within 3 weeks of the scheduled interruption, unless otherwise discussed with the Sponsor. The reason for interruption should be documented in the patient's study record.

Patients may continue on study treatment with either drug as monotherapy should they require discontinuation of one of the study drugs due to unacceptable toxicity or intolerance. Patients will continue to follow the study schedule and procedures, per protocol until discontinuation criteria is met for the second drug.



# 5.2.1.3 Dose Modification and toxicity management for immune-related AEs associated with pembrolizumab

AEs associated with pembrolizumab exposure may represent an immunologic etiology. These immune-related AEs (irAEs) may occur shortly after the first dose or several months after the last dose of pembrolizumab treatment and may affect more than one body system simultaneously. Therefore, early recognition and initiation of treatment is critical to reduce complications. Based on existing clinical trial data, most irAEs were reversible and could be managed with interruptions of pembrolizumab, administration of corticosteroids and/or other supportive care. For suspected irAEs, ensure adequate evaluation to confirm etiology or exclude other causes. Additional procedures or tests such as bronchoscopy, endoscopy, skin biopsy may be included as part of the evaluation. Based on the severity of irAEs, withhold or permanently discontinue pembrolizumab and administer corticosteroids. Dose modification and toxicity management guidelines for irAEs associated with pembrolizumab are provided in Table 3.

Table 3 Dose modification and toxicity management guidelines for immune-related AEs associated with pembrolizumab

#### **General instructions:**

- 1. Corticosteroid taper should be initiated upon AE improving to Grade 1 or less and continue to taper over at least 4 weeks.
- 2. For situations where pembrolizumab has been withheld, pembrolizumab can be resumed after AE has been reduced to Grade 1 or 0 and corticosteroid has been tapered. Pembrolizumab should be permanently discontinued if AE does not resolve within 12 weeks of last dose or corticosteroids cannot be reduced to ≤ 10 mg prednisone or equivalent per day within 12 weeks.
- **3.** For severe and life-threatening irAEs, IV corticosteroid should be initiated first followed by oral steroid. Other immunosuppressive treatment should be initiated if irAEs cannot be controlled by corticosteroids.

| Immune-related<br>AEs | Toxicity grade<br>or conditions<br>(CTCAEv5.0) | Action taken to pembrolizumab | irAE management<br>with<br>corticosteroid<br>and/or other<br>therapies | Monitor and follow-up |
|---|---|---|---|---|
| Pneumonitis | Grade 2 | Withhold | Administer corticosteroids (initial dose of | Monitor subjects for<br>signs and symptoms<br>of pneumonitis |
| | Grade 3 or 4, or recurrent grade 2 | Permanently discontinue | 1-2mg/kg<br>prednisone or<br>equivalent)<br>followed by<br>taper | Evaluate subjects with suspected pneumonitis with radiographic imaging and initiate corticosteroid |

17 v5 dated 10Dec2018



| Diarrhea / colitis | Grade 2 or 3 | Withhold | Administer corticosteroids (initial dose of 1-2mg/kg prednisone or equivalent) full and the | <ul> <li>treatment</li> <li>Add prophylactic antibiotics for opportunistic infections</li> <li>Monitor subjects for signs and symptoms of enterocolitis (i.e. diarrhea, abdominal pain, blood or mucus in stool with or</li> </ul> |
|---|---|---|---|---|
| | Grade 4 | Permanently discontinue | followed by taper taper (aa • S (c) S (c) (d) (d) (d) (d) (d) (d) (d) | Grade 2 diarrhea suspecting colitis should consider GI consultation and performing endoscopy to rule out colitis. |
| AST / ALT<br>elevation or<br>Increased<br>Bilirubin | Grade 2 | Withhold | Administer corticosteroids (initial dose of 0.5- 1mg/kg prednisone or equivalent) followed by taper | Monitor with liver function tests (consider weekly or more frequently until liver enzyme value returned to baseline or is stable |
| | Grade 3 or 4 | Permanently discontinue | Administer corticosteroids (initial dose of 1-2mg/kg prednisone or equivalent) followed by taper | |



| Type 1 diabetes<br>mellitus (T1DM)<br>or Hyperglycemia | Newly onset<br>T1DM or<br>Grade 3 or 4<br>hyperglycemia<br>associated with<br>evidence of β-cell<br>failure | Withhold | <ul> <li>Initiate insulin replacement therapy for subjects with T1DM</li> <li>Administer antihyperglycemic in subjects with hyperglycemia</li> </ul> | • | Monitor subjects for<br>hyperglycemia or<br>other signs and<br>symptoms of<br>diabetes. |
|---|---|---|---|---|---|
| Hypophysitis | Grade 2 | Withhold | Administer corticosteroids and initiate | • | Monitor for signs and symptoms of hypophysitis |
| | Grade 3 or 4 | Withhold or<br>permanently<br>discontinue <sup>1</sup> | hormonal<br>replacements as<br>clinically<br>indicated. | | (including<br>hypopituitarism and<br>adrenal insufficiency) |
| Hyperthyroidism | Grade 2 | Continue | Treat with non-<br>selective beta-<br>blockers (e.g. | • | Monitor for signs and symptoms of thyroid disorders. |
| | Grade 3 or 4 | Withhold or<br>Permanently<br>discontinue <sup>1</sup> | propranolol) or<br>thionamides as<br>appropriate | | |
| Hypothyroidism | Grade 2-4 | Continue | Initiate thyroid<br>replacement<br>hormones (e.g.<br>levothyroxine<br>or<br>liothyroinine)<br>per standard of<br>care | • | Monitor for signs and symptoms of thyroid disorders. |
| Nephritis and renal dysfunction | Grade 2 | Withhold | Administer corticosteroids | • | Monitor changes of renal function |
| , | Grade 3 or 4 | Permanently discontinue | (prednisone 1-<br>2mg/kg or<br>equivalent)<br>followed by<br>taper. | | |
| All Other<br>immune-related<br>AEs | Grade 3, or intolerable/ persistent Grade 2 | Withhold | Based on<br>severity of AE<br>administer<br>corticosteroids | • | Ensure adequate evaluation to confirm etiology or exclude other causes |
| | Grade 4 or recurrent Grade 3 | Permanently discontinue | | | |



#### **NOTES:**

- 1. Withholding or permanently discontinuing pembrolizumab is at the discretion of the investigator or treating physician.
- 2. For subjects with Grade 3 or 4 immune-related endocrinopathy where withhold of pembrolizumab is required, pembrolizumab may be resumed when AE resolves to ≤ Grade 2 and is controlled with hormonal replacement therapy or achieved metabolic control (in case of T1DM)

# 5.2.1.3 Dose modification and toxicity management of infusion-reactions related to pembrolizumab

Pembrolizumab may cause severe or life threatening infusion-reactions including severe hypersensitivity or anaphylaxis. Signs and symptoms usually develop during or shortly after drug infusion and generally resolve completely within 24 hours of completion of infusion. Dose modification and toxicity management guidelines on pembrolizumab associated infusion reaction are provided in Table 4.

Table 4 Pembrolizumab Infusion Reaction Dose modification and Treatment Guidelines

| NCI CTCAE Grade | Treatment | Premedication at<br>Subsequent Dosing |
|---|---|---|
| Grade 1 Mild reaction; infusion interruption not indicated; intervention not indicated | Increase monitoring of vital signs as medically indicated until the subject is deemed medically stable in the opinion of the investigator. | None |



| Grade 2 | Stop Infusion. | Subject may be premedicated |
|---|---|---|
| Requires therapy or | Additional appropriate medical therapy may | 1.5h (± 30 minutes) prior to |
| infusion interruption but | include but is not limited to: | infusion of pembrolizumab |
| responds promptly to | IV fluids | with: |
| symptomatic treatment | Antihistamines | Diphenhydramine 50 mg po |
| (e.g., antihistamines, | NSAIDs | (or equivalent dose of |
| NSAIDs, narcotics, IV | Acetaminophen | antihistamine). |
| fluids); prophylactic | Narcotics | Acetaminophen 500-1000 mg |
| medications indicated | Increase monitoring of vital signs as medically | po (or equivalent dose of |
| for ≤24 hrs | indicated until the subject is deemed medically | analgesic). |
| | stable in the opinion of the investigator. | unuigesie). |
| | If symptoms resolve within 1 hour of stopping | |
| | drug infusion, the infusion may be restarted at | |
| | 50% of the original infusion rate (e.g. from 100 | |
| | mL/hr to 50 mL/hr). Otherwise dosing will be | |
| | held until symptoms resolve and the subject | |
| | should be premedicated for the next scheduled | |
| | dose. | |
| | Subjects who develop Grade 2 toxicity despite | |
| | adequate premedication should be permanently | |
| | discontinued from further study drug | |
| | treatment | |
| Grades 3 or 4 | Stop Infusion. | No subsequent dosing |
| Grade 3: | Additional appropriate medical therapy may | |
| Prolonged (i.e., not | include but is not limited to: | |
| rapidly responsive to | Epinephrine** | |
| symptomatic medication | IV fluids | |
| and/or brief interruption | Antihistamines | |
| of infusion); recurrence | NSAIDs | |
| of symptoms following | Acetaminophen | |
| initial improvement; | Narcotics | |
| hospitalization indicated | Oxygen | |
| for other clinical | Pressors | |
| sequelae (e.g., renal | Corticosteroids | |
| impairment, pulmonary | Increase monitoring of vital signs as medically | |
| infiltrates) | indicated until the subject is deemed medically | |
| Grade 4: | stable in the opinion of the investigator. | |
| Life-threatening; | Hospitalization may be indicated. | |
| pressor or ventilatory | **In cases of anaphylaxis, epinephrine should be | |
| support indicated | used immediately. | |
| | Subject is permanently discontinued from | |
| | further study drug treatment. | |
| Appropriate resuscitation equipment should be available at the bedside and a physician readily available during the period of | | |

Appropriate resuscitation equipment should be available at the bedside and a physician readily available during the period of drug administration.

For further information, please refer to the Common Terminology Criteria for Adverse Events v5.0 (CTCAE) at http://ctep.cancer.gov

# 5.2.1.3 Dose Modification and toxicity management for AEs associated with lenvatinib



# Hypertension

- Assess blood pressure prior to and periodically during treatment. Initiate or adjust medical management to control blood pressure prior to and during treatment.
- Withhold lenvatinib for Grade 3 hypertension that persists despite optimal antihypertensive therapy; resume at a reduced dose (see Table 1) when hypertension is controlled at less than or equal to Grade 2.
- Discontinue lenvatinib for life-threatening hypertension.

# Cardiac dysfunction or hemorrhage

- Discontinue for a Grade 4 event.
- Withhold lenvatinib for development of Grade 3 event until improved to Grade 0 or 1 or baseline.
- Either resume at a reduced dose (see Table 1) or discontinue lenvatinib depending on the severity and persistence of the adverse event.

#### Arterial thrombotic event

• Discontinue lenvatinib following an arterial thrombotic event.

# Renal failure and impairment or hepatotoxicity

- Withhold lenvatinib for development of Grade 3 or 4 renal failure/impairment or hepatotoxicity until resolved to Grade 0 to 1 or baseline.
- Either resume at a reduced dose (see Table 1) or discontinue lenvatinib depending on the severity and persistence of renal impairment or hepatotoxicity.
- Discontinue lenvatinib for hepatic failure.

#### Proteinuria

- Withhold lenvatinib for ≥2 grams of proteinuria/24 hours.
- Resume at a reduced dose (see Table 1) when proteinuria is <2 gm/24 hours.
- Discontinue lenvatinib for nephrotic syndrome.

# Gastrointestinal perforation or fistula formation



• Discontinue lenvatinib in patients who develop gastrointestinal perforation or lifethreatening fistula.

# QT prolongation

- Withhold lenvatinib for the development of Grade 3 or greater QT interval prolongation.
- Resume lenvatinib at a reduced dose (see Table 1) when QT prolongation resolves to Grade 0 or 1 or baseline.

Reversible posterior leukoencephalopathy syndrome (RPLS)

- Withhold for RPLS until fully resolved.
- Upon resolution, resume at a reduced dose or discontinue lenvatinib depending on the severity and persistence of neurologic symptoms.

Manage other adverse reactions according to the instructions in Table 5. Based on the absence of clinical experience, there are no recommendations on resumption of dosing in patients with Grade 4 clinical adverse reactions that resolve.



Table 4 Recommended Dose Modifications for Persistent and Intolerable Grade 2 or Grade 3 Adverse Reactions or Grade 4 Laboratory Abnormalities<sup>a</sup>

| Adverse Reaction | Modification | Adjusted Dose <sup>b</sup> |
|---|---|---|
| First occurrence | Interrupt until resolved to | 20 mg (two 10 mg capsules) |
| Thist occurrence | Grade 0-1 or baseline | orally once daily |
| Second occurrence <sup>c</sup> | Interrupt until resolved to Grade 0-1 or baseline | 14 mg (one 10 mg capsule plus<br>one 4 mg capsule) orally once<br>daily |
| Third occurrence <sup>c</sup> | Interrupt until resolved to Grade 0-1 or baseline | 10 mg (one 10 mg capsule) orally once daily |

- a. Initiate medical management for nausea, vomiting, or diarrhea prior to interruption or dose reduction of lenvatinib
- b. Reduce dose in succession based on the previous dose level (24 mg, 20 mg, or 14 mg per day)
- c. Refers to the same or a different adverse reaction that requires dose modification

### **5.2.2** Timing of Dose Administration

Trial treatment should be administered on Day 1 of each cycle after all procedures/assessments have been completed as detailed on the Trial Flow Chart (Section 6.0). Trial treatment may be administered up to 3 days before or after the scheduled Day 1 of each cycle due to administrative reasons.

All trial treatments will be administered on an outpatient basis.

Pembrolizumab 200 mg will be administered as a 30 minute IV infusion every 3 weeks. Sites should make every effort to target infusion timing to be as close to 30 minutes as possible. However, given the variability of infusion pumps from site to site, a window of -5 minutes and +10 minutes is permitted (i.e., infusion time is 30 minutes: -5 min/+10 min).

Lenvatinib 24 mg will be administered orally and provided in 10mg and 4mg capsules (supplied in cartons of 6 cards; each card is a 5-day blister card), taken daily with or without food. Lenvatinib should be taken at the same time each day. If a dose is missed and cannot be taken within 12 hours, patients should skip that dose and take the next dose at the usual time of administration. Patients will be required to maintain documentation of all dose administrations on a pill diary each cycle.



The Pharmacy Manual contains specific instructions for the preparation of the pembrolizumab infusion fluid and administration of infusion solution. Lenvatinib will be dispensed and handled according to the FDA approved package insert.

## 5.2.3 Trial Blinding/Masking

This is an open-label trial; therefore, the Sponsor, investigator and subject will know the treatment administered.

# 5.3 Concomitant Medications/Vaccinations (allowed & prohibited)

Medications or vaccinations specifically prohibited in the exclusion criteria are not allowed during the ongoing trial. If there is a clinical indication for one of these or other medications or vaccinations specifically prohibited during the trial, discontinuation from trial therapy or vaccination may be required. The investigator should discuss any questions regarding this with the Merck Clinical team. The final decision on any supportive therapy or vaccination rests with the investigator and/or the subject's primary physician.

# 5.3.1 Acceptable Concomitant Medications

All treatments that the investigator considers necessary for a subject's welfare may be administered at the discretion of the investigator in keeping with the community standards of medical care. All concomitant medication will be recorded on the case report form (CRF) including all prescription, over-the-counter (OTC), herbal supplements, and IV medications and fluids. If changes occur during the trial period, documentation of drug dosage, frequency, route, and date may also be included on the CRF.

All concomitant medications received within 28 days before the first dose of trial treatment and 30 days after the last dose of trial treatment should be recorded. Concomitant medications administered after 30 days after the last dose of trial treatment should be recorded for SAEs and ECIs as defined in Section 7.2. Somatostatin analogs (octreotide and lanreotide) are rarely used in patients with poorly differentiated/high grade neuroendocrine cancers, but are allowed if needed for control of hormonal syndromes.

### **5.3.2** Prohibited Concomitant Medications

Subjects are prohibited from receiving the following therapies during the Screening and Treatment Phase (including retreatment for post-complete response relapse) of this trial:

- Antineoplastic systemic chemotherapy or biological therapy
- Immunotherapy not specified in this protocol
- Chemotherapy not specified in this protocol



- Investigational agents other than pembrolizumab
- Radiation therapy
  - Note: Radiation therapy to a symptomatic solitary lesion or to the brain may be allowed at the investigator's discretion.
- Live vaccines within 30 days prior to the first dose of trial treatment and while participating in the trial. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, BCG, and typhoid vaccine.
- Systemic glucocorticoids for any purpose other than to modulate symptoms from an event of clinical interest of suspected immunologic etiology. The use of physiologic doses of corticosteroids may be approved after consultation with the Sponsor.
- Strong CYP3A, P-glycoprotein (P-gp), and breast cancer resistance protein (BCRP) inhibitors and CYP3A and P-gp inducers are not prohibited, but should be avoided while on study therapy.
- Grapefruit, grapefruit juice, or Seville oranges

Subjects who, in the assessment by the investigator, require the use of any of the aforementioned treatments for clinical management should be removed from the trial. Subjects may receive other medications that the investigator deems to be medically necessary.

The Exclusion Criteria describes other medications which are prohibited in this trial.

There are no prohibited therapies during the Post-Treatment Follow-up Phase.

# 5.4 Diet/Activity/Other Considerations

#### **5.4.1** Diet

Subjects should maintain a normal diet unless modifications are required to manage an AE such as diarrhea, nausea or vomiting.

# 5.4.2 Contraception

The study drugs may have adverse effects on a fetus in utero. Furthermore, it is not known if these drugs havetransient adverse effects on the composition of sperm.

For this trial, male subjects will be considered to be of non-reproductive potential if they have azoospermia (whether due to having had a vasectomy or due to an underlying medical condition).



Female subjects will be considered of non-reproductive potential if they are either:

(1) postmenopausal (defined as at least 12 months with no menses without an alternative medical cause; in women < 45 years of age a high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. In the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.);

OR

(2) have had a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy or bilateral tubal ligation/occlusion, at least 6 weeks prior to screening;

OR

(3) has a congenital or acquired condition that prevents childbearing.

Female and male subjects of reproductive potential must agree to avoid becoming pregnant or impregnating a partner, respectively, while receiving study drug and for 120 days after the last dose of study drug by complying with one of the following:

(1) practice abstinence<sup>†</sup> from heterosexual activity;

OR

(2) use (or have their partner use) acceptable contraception during heterosexual activity.

Acceptable methods of contraception are<sup>‡</sup>:

Single method (one of the following is acceptable):

- intrauterine device (IUD)
- vasectomy of a female subject's male partner
- contraceptive rod implanted into the skin

Combination method (requires use of two of the following):



- diaphragm with spermicide (cannot be used in conjunction with cervical cap/spermicide)
- cervical cap with spermicide (nulliparous women only)
- contraceptive sponge (nulliparous women only)
- male condom or female condom (cannot be used together)
- hormonal contraceptive: oral contraceptive pill (estrogen/progestin pill or progestinonly pill), contraceptive skin patch, vaginal contraceptive ring, or subcutaneous contraceptive injection

†Abstinence (relative to heterosexual activity) can be used as the sole method of contraception if it is consistently employed as the subject's preferred and usual lifestyle and if considered acceptable by local regulatory agencies and ERCs/IRBs. Periodic abstinence (e.g., calendar, ovulation, sympto-thermal, post-ovulation methods, etc.) and withdrawal are not acceptable methods of contraception.

‡If a contraceptive method listed above is restricted by local regulations/guidelines, then it does not qualify as an acceptable method of contraception for subjects participating at sites in this country/region.

Subjects should be informed that taking the study medication may involve unknown risks to the fetus (unborn baby) if pregnancy were to occur during the study. In order to participate in the study subjects of childbearing potential must adhere to the contraception requirement (described above) from the day of study medication initiation (or 14 days prior to the initiation of study medication for oral contraception) throughout the study period up to 120 days after the last dose of trial therapy. If there is any question that a subject of childbearing potential will not reliably comply with the requirements for contraception, that subject should not be entered into the study.

### 5.4.3 Use in Pregnancy

If a subject inadvertently becomes pregnant while on study treatment, the subject will immediately be removed from the study. The site will contact the subject at least monthly and document the subject's status until the pregnancy has been completed or terminated. The outcome of the pregnancy will be reported to the Sponsor and to Merck without delay and



within 24 hours to the Sponsor and within 2 working days to Merck if the outcome is a serious adverse experience (e.g., death, abortion, congenital anomaly, or other disabling or life-threatening complication to the mother or newborn).

The study investigator will make every effort to obtain permission to follow the outcome of the pregnancy and report the condition of the fetus or newborn to the Sponsor. If a male subject impregnates his female partner the study personnel at the site must be informed immediately and the pregnancy reported to the Sponsor and to Merck and followed as described above and in Section 7.2.2.

# 5.4.4 Use in Nursing Women

It is unknown whether pembrolizumab and/or lenvatinib are excreted in human milk. Since many drugs are excreted in human milk, and because of the potential for serious adverse reactions in the nursing infant, subjects who are breast-feeding are not eligible for enrollment.

## 5.5 Subject Withdrawal/Discontinuation Criteria

Subjects may withdraw consent at any time for any reason or be dropped from the trial at the discretion of the investigator should any untoward effect occur. In addition, a subject may be withdrawn by the investigator or the Sponsor if enrollment into the trial is inappropriate, the trial plan is violated, or for administrative and/or other safety reasons. Specific details regarding discontinuation or withdrawal are provided in Section 7.1.3 – Other Procedures.

A subject must be discontinued from the trial for any of the following reasons:

- The subject or legal representative (such as a parent or legal guardian) withdraws consent.
- Confirmed radiographic disease progression
- Unacceptable adverse experiences as described in Section 5.2.1.2
- Intercurrent illness that prevents further administration of treatment
- Investigator's decision to withdraw the subject
- The subject has a confirmed positive serum pregnancy test
- Noncompliance with trial treatment or procedure requirements
- The subject is lost to follow-up



- Completed 24 months of uninterrupted treatment with pembrolizumab or 35 administrations of study medication, whichever is later.
- Administrative reasons

The End of Treatment and Follow-up visit procedures are listed in Section 6 (Protocol Flow Chart) and Section 7.1.4 (Visit Requirements). After the end of treatment, each subject will be followed for 30 days for adverse event monitoring (serious adverse events will be collected for 90 days after the end of treatment as described in Section 7.2.3.1). Subjects who discontinue for reasons other than progressive disease will have post-treatment follow-up for disease status until disease progression, initiating a non-study cancer treatment, withdrawing consent or becoming lost to follow-up. After documented disease progression each subject will be followed by telephone for overall survival until death, withdrawal of consent, or the end of the study, whichever occurs first.

# 5.6 Subject Replacement Strategy

Subjects who enroll but do not receive first dose of trial drug will be replaced

# 5.7 Clinical Criteria for Early Trial Termination

Early trial termination will be the result of the criteria specified below:

- 1. Quality or quantity of data recording is inaccurate or incomplete
- 2. Poor adherence to protocol and regulatory requirements
- 3. Incidence or severity of adverse drug reaction in this or other studies indicates a potential health hazard to subjects
- 4. Plans to modify or discontinue the development of the study drug

In the event of Merck decision to no longer supply study drugs, ample notification will be provided so that appropriate adjustments to subject treatment can be made.

# 6.0 TRIAL FLOW CHART

# 6.1 Study Flow Chart

| Trial Period: | Screenin | ng Phase | Treatment Cycles <sup>a</sup> | | | | | | | End of<br>Treatment | Post-Treatment | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Pre- | Main<br>Study | | | | | To be repeated beyond 8 cycles | | | | | | | Survival |
| Treatment Cycle/Title: | screening<br>(Visit 1) | Screening<br>(Visit 2) | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | Discon | Safety<br>Follow-up | Follow Up<br>Visits <sup>c</sup> | Follow-<br>Up |
| Scheduling Window (Days): | -42 to -1 | -14 to -1 | | ± 3 | ± 3 | ± 3 | ± 3 | ± 3 | ± 3 | ± 3 | At time of Discon | 30 days<br>post<br>discon | Every 9<br>weeks post<br>discon | Every<br>12<br>weeks |
| Administrative Procedures | | | | L | L | <u>L</u> | L | • | | | | | <u> </u> | - |
| Informed Consent | X | | | | | | | | | | | | | |
| Inclusion/Exclusion Criteria | | X | | | | | | | | | | | | |
| Demographics and Medical History | | X | | | | | | | | | | | | |
| Prior and Concomitant Medication Review | | X | X | X | X | X | X | X | X | X | | | | |
| Study drug Administration | | | X | X | X | X | X | X | X | X | | | | |
| Survival Status | | | | | | | | | | | | | | X |
| Clinical Procedures/Assessments | | | | , | , | | , | | | | | • | | |
| Review Adverse Events | | X | X | X | X | X | X | X | X | X | X | X | | |
| Full Physical Examination | | X | | | | | | | | | X | | | |
| Directed Physical Examination | | | X | X | X | X | X | X | X | X | | | | |
| Vital Signs and Weight | | X | X | X | X | X | X | X | X | X | X | X | | |
| ECOG Performance Status | | X | X | X | X | X | X | X | X | X | X | X | | |
| Electrocardiogram | | X | | | | Xa | | | | | | | | |
| Laboratory Procedures/Assessments: analy | ysis perforn | · · | AL lab | orator | y | | | | | | | | | |
| Pregnancy Test –Serum β-HCG | | Xb | | | | | | | | | | | | |
| PT/INR and aPTT | | X | | | | | | | | | | | | |
| CBC with Differential | | X | X | X | X | X | X | X | X | X | X | X | | |
| Comprehensive Serum Chemistry Panel | | X | X | X | X | X | X | X | X | X | X | X | | |

| Trial Period: | Screenir | ng Phase | Treatment Cycles <sup>a</sup> | | | | | | | End of<br>Treatment | Post-Treatment | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Pre- | Main<br>Study | | | | | To be repeated beyond 8 cycles | | | | | | Survival | |
| Treatment Cycle/Title: | screening<br>(Visit 1) | Screening (Visit 2) | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | Discon | Safety<br>Follow-up | Follow Up<br>Visits <sup>c</sup> | Follow-<br>Up |
| Scheduling Window (Days): | -42 to -1 | -14 to -1 | | ± 3 | ± 3 | ± 3 | ± 3 | ± 3 | ± 3 | ± 3 | At time of Discon | 30 days<br>post<br>discon | Every 9<br>weeks post<br>discon | Every<br>12<br>weeks |
| Urinalysis | | X <sup>c</sup> | X | | X | | X | | X | | | X | | |
| T3, FT4 and TSH | | X <sup>c</sup> | | X | | X | | X | | X | | X | | |
| Efficacy Measurements | | | | | | | | | | | | | | |
| Tumor Imaging | | $X^{f}$ | | | $X^d$ | | | X | | | | | X | |
| Archival Tissue Collection/Correlative Studies Blood | | | | | | | | | | | | | | |
| Archival Tissue Collection | X <sup>e</sup> | | | | | | | | | | | | | |

- a. ECG at baseline and at each restaging assessment for patients that are symptomatic or have QTcF at baseline of >450ms
- b. For women of reproductive potential, a serum pregnancy test should be performed within 72 hours prior to first dose of trial treatment and repeated at each restaging assessment.
- c. Every other cycle (including beyond cycle 8). Add on 24-hour urine protein for any visit with urine protein 1+ (>30mg/dL)
- d. The first on-study imaging time point will be at 9 weeks (+/- 7 days) after the date of cycle 1 day 1, then every 9 weeks (+/- 7 days) thereafter. After 12 months, imaging frequency should be reduced to every 12 weeks (+/- 7 days). Imaging timing should follow calendar days and should not be adjusted for delays in cycle starts.
- e. Archival tumor collection can be performed at any time during the study and is not a prerequisite for enrollment or initiation of treatment
- f. Tumor imaging for screening may be at day -28 to -1

### 7.0 TRIAL PROCEDURES

#### 7.1 Trial Procedures

The Trial Flow Chart - Section 6.0 summarizes the trial procedures to be performed at each visit. Individual trial procedures are described in detail below. It may be necessary to perform these procedures at unscheduled time points if deemed clinically necessary by the investigator.

Furthermore, additional evaluations/testing may be deemed necessary by the Sponsor and/or Merck for reasons related to subject safety. In some cases, such evaluation/testing may be potentially sensitive in nature (e.g., HIV, Hepatitis C, etc.), and thus local regulations may require that additional informed consent be obtained from the subject. In these cases, such evaluations/testing will be performed in accordance with those regulations.

#### 7.1.1 Administrative Procedures

#### 7.1.1.1 Informed Consent

The Investigator must obtain documented consent from each potential subject prior to participating in a clinical trial.

### 7.1.1.1.1 General Informed Consent

Consent must be documented by the subject's dated signature or by the subject's legally acceptable representative's dated signature on a consent form along with the dated signature of the person conducting the consent discussion.

A copy of the signed and dated consent form should be given to the subject before participation in the trial.

The initial informed consent form, any subsequent revised written informed consent form and any written information provided to the subject must receive the IRB/ERC's approval/favorable opinion in advance of use. The subject or his/her legally acceptable representative should be informed in a timely manner if new information becomes available that may be relevant to the subject's willingness to continue participation in the trial. The communication of this information will be provided and documented via a revised consent form or addendum to the original consent form that captures the subject's dated signature or by the subject's legally acceptable representative's dated signature.

Specifics about a trial and the trial population will be added to the consent form template at the protocol level.

The informed consent will adhere to IRB/ERC requirements, applicable laws and regulations and Sponsor requirements.

### 7.1.1.2 Inclusion/Exclusion Criteria

All inclusion and exclusion criteria will be reviewed by the investigator or qualified designee to ensure that the subject qualifies for the trial.

# 7.1.1.3 Medical History

A medical history will be obtained by the investigator or qualified designee. Medical history will include all active conditions, and any condition diagnosed within the prior 10 years that are considered to be clinically significant by the Investigator. Details regarding the disease for which the subject has enrolled in this study will be recorded separately and not listed as medical history.

#### 7.1.1.4 Prior and Concomitant Medications Review

### 7.1.1.4.1 Prior Medications

The investigator or qualified designee will review prior medication use, including any protocol-specified washout requirement, and record prior medication taken by the subject within 28 days before starting the trial. Treatment for the disease for which the subject has enrolled in this study will be recorded separately and not listed as a prior medication.

### 7.1.1.4.2 Concomitant Medications

The investigator or qualified designee will record medication, if any, taken by the subject during the trial during all visits. All medications related to reportable SAEs and ECIs should be recorded as defined in Section 7.2.

#### 7.1.1.5 Disease Details and Treatments

### 7.1.1.5.1 Disease Details

The investigator or qualified designee will obtain prior and current details regarding disease status.

# 7.1.1.5.2 Prior Treatment Details

The investigator or qualified designee will review all prior cancer treatments including systemic treatments, radiation and surgeries.

# 7.1.1.5.3 Subsequent Anti-Cancer Therapy Status

The investigator or qualified designee will review all new anti-neoplastic therapy initiated after the last dose of trial treatment. If a subject initiates a new anti-cancer therapy within 30 days after the last dose of trial treatment, the 30 day Safety Follow-up visit must occur before the first dose of the new therapy. Once new anti-cancer therapy has been initiated the subject will move into survival follow-up.

### 7.1.2 Clinical Procedures/Assessments

# 7.1.2.1 Adverse Event (AE) Monitoring

The investigator or qualified designee will assess each subject to evaluate for potential new or worsening AEs as specified in the Trial Flow Chart and more frequently if clinically indicated. Adverse experiences will be graded and recorded throughout the study and during the follow-up period according to NCI CTCAE Version 5.0 (see Section 11.2). Toxicities will be characterized in terms regarding seriousness, causality, toxicity grading, and action taken with regard to trial treatment.

Please refer to section 7.2 for detailed information regarding the assessment and recording of AEs.

# 7.1.2.2 Full Physical Exam

The investigator or qualified designee will perform a complete physical exam during the screening period. Clinically significant abnormal findings should be recorded as medical history. A full physical exam should be performed during screening,

# 7.1.2.3 Directed Physical Exam

For cycles that do not require a full physical exam per the Trial Flow Chart, the investigator or qualified designee will perform a directed physical exam as clinically indicated prior to trial treatment administration.

# **7.1.2.4** Vital Signs

The investigator or qualified designee will take vital signs at screening, prior to the administration of each dose of trial treatment and at treatment discontinuation as specified in the Trial Flow Chart (Section 6.0). Vital signs should include temperature, pulse, respiratory rate, weight and blood pressure. Height will be measured at screening only.

# 7.1.2.5 Eastern Cooperative Oncology Group (ECOG) Performance Scale

The investigator or qualified designee will assess ECOG status (see Section 11.1) at screening, prior to the administration of each dose of trial treatment and discontinuation of trial treatment as specified in the Trial Flow Chart.

# 7.1.2.6 Tumor Imaging and Assessment of Disease

Tumor imaging of the chest, abdomen and pelvis should be performed by computed tomography (CT) with iv contrast. An alternative is an MRI of the abdomen/pelvis with iv contrast and a chest CT (with or without iv contrast).
# 7.1.2.7 Initial Tumor Imaging

Initial tumor imaging must be performed within 28 days prior to the first dose of trial treatment. Scans performed as part of routine clinical management are acceptable for use as the screening scan if they are of diagnostic quality and performed within 28 days prior to the first dose of trial treatment. The same imaging technique should be used for a given subject throughout the trial.

## 7.1.2.8 Tumor imaging During Trial

The first imaging assessment during treatment should be performed at 9 weeks ( $63 \pm 7$  days) from Cycle 1, Day 1. Subsequent imaging should initially be performed every 9 weeks ( $63 \pm 7$  days) or more frequently, if clinically indicated. After the first 12 months on trial therapy, the imaging interval should be increased to every 12 weeks ( $84 \pm 7$  days). Imaging timing should follow calendar days and should not be adjusted for delays in cycle starts. Imaging should continue to be performed until disease progression, the start of new anti-cancer treatment, withdrawal of consent, death, or notification by the Sponsor, whichever occurs first.

Per RECIST 1.1, PRs and CRs should be confirmed by a repeat tumor imaging assessment not less than 4 weeks from the date the response was first documented. The tumor imaging for confirmation of response may be performed at the earliest 4 weeks after the first indication of response, or at the next scheduled scan (i.e., 9 weeks later). Subjects will then return to regular scheduled imaging every 9 weeks, starting with the next scheduled imaging time point. Subjects who obtain a confirmation scan do not need to undergo the next scheduled tumor imaging if it is < 4 weeks later; tumor imaging may resume at the subsequent scheduled imaging time point.

## 7.1.2.9 Tumor Tissue Collection

Archival tissue will be obtained, if available, to assess for PD-L1 expression and MMR status. Availability of archival tissue will not be required for trial enrollment.

## 7.1.3 Laboratory Procedures/Assessments

Details regarding specific laboratory procedures/assessments to be performed in this trial are provided below (Laboratory Safety Evaluations (Hematology, Chemistry and Urinalysis)

Laboratory tests for hematology, chemistry, urinalysis, and others are specified in Table 7.

Table 6: Laboratory Tests

| Hematology | Chemistry | Urinalysis | Other |
|---|---|---|---|
| Hematocrit | Albumin | Blood | Serum β-human chorionic gonadotropin† |
| Hemoglobin | Alkaline phosphatase | Glucose | (β-hCG)† |
| Platelet count | Alanine aminotransferase (ALT) | Protein | PT (INR) |
| WBC (total and differential) | Aspartate aminotransferase (AST) | Specific gravity | aPTT |
| Red Blood Cell Count | Carbon Dioxide | Microscopic exam (If abnormal) | Total thriiodothyronine (T3) |
| Absolute Neutrophil Count | (CO <sub>2</sub> or biocarbonate) | results are noted | Free tyroxine (T4) |
| Absolute Lymphocyte Count | Calcium | | Thyroid stimulating hormone (TSH) |
| | Chloride | | |
| | Glucose | | |
| | Potassium | | |
| | Sodium | | |
| | Total Bilirubin | | |
| | Total protein | | |
| | Blood Urea Nitrogen | | |
| † Perform on women of childbea | ring potential only. | , | ' |

Laboratory tests for screening should be performed within 28 days prior to the first dose of treatment. After Cycle 1, pre-dose laboratory procedures can be conducted up to 72 hours prior to dosing. Results must be reviewed by the investigator or qualified designee and found to be acceptable prior to each dose of trial treatment.

### 7.1.4 Other Procedures

## 7.1.4.1 Withdrawal/Discontinuation

When a subject discontinues/withdraws prior to trial completion, all applicable activities scheduled for the final trial visit should be performed at the time of discontinuation. Any adverse events which are present at the time of discontinuation/withdrawal should be followed in accordance with the safety requirements outlined in Section 7.2 - Assessing and Recording Adverse Events. Subjects who a) attain a CR or b) complete 24 months of treatment with pembrolizumab may discontinue treatment with the option of restarting treatment if they meet the criteria specified in Section 7.1.5.5. After discontinuing treatment following assessment of CR, these subjects should return to the site for a Safety Follow-up Visit (described in Section 7.1.5.3.1) and then proceed to the Follow-Up Period of the study (described in Section 7.1.5.4).

# 7.1.5 Visit Requirements

Visit requirements are outlined in Section 6.0 - Trial Flow Chart. Specific procedure-related details are provided above in Section 7.1 - Trial Procedures.

## **7.1.5.1** Screening

Within 42 days prior to enrollment, potential subjects will be evaluated to determine if they fulfill the entry requirements as set forth in section 5.1. Screening procedures may be repeated.

Imaging for baseline tumor assessment, laboratory tests and ECOG status are to be performed within 28 days prior to the first dose of trial treatment

For women of reproductive potential, a serum pregnancy test will be performed 72 hours prior to the first dose of trial treatment.

## 7.1.5.2 Treatment Period

Visit requirements are outlined in section 6.0 – Trial Flow Chart. A window of  $\pm$  days is permitted for tests and trial drug infusion

### 7.1.5.3 Post-Treatment Visits

## 7.1.5.3.1 Safety Follow-Up Visit

The mandatory Safety Follow-Up Visit should be conducted approximately 30 days after the last dose of trial treatment or before the initiation of a new anti-cancer treatment, whichever comes first. All AEs that occur prior to the Safety Follow-Up Visit should be recorded. Subjects with an AE of Grade > 1 will be followed until the resolution of the AE to Grade 0-1 or until the beginning of a new anti-neoplastic therapy, whichever occurs first. SAEs that occur within 90 days of the end of treatment or before initiation of a new anti-cancer treatment should also be followed and recorded. Subjects who are eligible for retreatment with pembrolizumab (as described in Section 7.1.5.5) may have up to two safety follow-up visits, one after the Treatment Period and one after the Second Course Phase.

## 7.1.5.4 Follow-up Visits

Subjects who discontinue trial treatment for a reason other than disease progression will move into the Follow-Up Phase and should be assessed every 9 (+/- 7 days) weeks with radiologic imaging to monitor disease status. Every effort should be made to collect information regarding disease status until the start of new anti-neoplastic therapy, disease progression, death, end of the study or if the subject begins retreatment with pembrolizumab as detailed in Section 7.1.5.5. Information regarding post-study anti-neoplastic treatment will be collected if new treatment is initiated.

# 7.1.5.4.1 Survival Follow-up

Once a subject experiences confirmed disease progression or starts a new anti-cancer therapy, the subject moves into the survival follow-up phase and should be contacted by telephone every 12 weeks to assess for survival status until death, withdrawal of consent, or the end of the study, whichever occurs first.

## 7.2 Assessing and Recording Adverse Events

An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Merck's product, is also an adverse event.

Changes resulting from normal growth and development that do not vary significantly in frequency or severity from expected levels are not to be considered adverse events. Examples of this may include, but are not limited to, teething, typical crying in infants and children and onset of menses or menopause occurring at a physiologically appropriate time.

Merck product includes any pharmaceutical product, biological product, device, diagnostic agent or protocol-specified procedure, whether investigational (including placebo or active comparator medication) or marketed, manufactured by, licensed by, provided by or distributed by Merck for human use.

Adverse events may occur during the course of the use of Merck product in clinical trials, or as prescribed in clinical practice, from overdose (whether accidental or intentional), from abuse and from withdrawal.

Progression of the cancer under study is not considered an adverse event.

All adverse events that occur after the consent form is signed but before treatment allocation/randomization must be reported by the investigator if they cause the subject to be excluded from the trial, or are the result of a protocol-specified intervention, including but not limited to washout or discontinuation of usual therapy, diet, placebo treatment or a procedure.

From the time of treatment allocation/randomization through 30 days following cessation of treatment, all adverse events must be reported by the investigator. Such events will be recorded at each examination on the Adverse Event case report forms/worksheets. The reporting timeframe for adverse events meeting any serious criteria is described in section 7.2.3.1. The investigator will make every attempt to follow all subjects with non-serious adverse events for outcome.

Laboratory tests and vital signs which fall out of normal range will only be reported as adverse events if considered clinically significant by the investigator.

# 7.2.1 Definition of an Overdose for This Protocol and Reporting of Overdose to the Sponsor and to Merck

For purposes of this trial, an overdose of pembrolizumab will be defined as any dose of 1,000 mg or greater (≥5 times the indicated dose). An overdose of lenvatinib will be defined as any dose of 120 mg or greater (≥5 times the indicated dose). No specific information is available on the treatment of overdose of pembrolizumab or lenvatinib. Appropriate supportive treatment should be provided if clinically indicated. In the event of overdose, the subject should be observed closely for signs of toxicity. Appropriate supportive treatment should be provided if clinically indicated.

If an adverse event(s) is associated with ("results from") the overdose of a Merck product, the adverse event(s) is reported as a serious adverse event, even if no other seriousness criteria are met.

If a dose of Merck's product meeting the protocol definition of overdose is taken without any associated clinical symptoms or abnormal laboratory results, the overdose is reported as a non-serious Event of Clinical Interest (ECI), using the terminology "accidental or intentional overdose without adverse effect."

All reports of overdose with and without an adverse event must be reported within 24 hours to the Sponsor and within 2 working days hours to Merck Global Safety. (Attn: Worldwide Product Safety; FAX 215 993-1220)

# 7.2.2 Reporting of Pregnancy and Lactation to the Sponsor and to Merck

Although pregnancy and lactation are not considered adverse events, it is the responsibility of investigators or their designees to report any pregnancy or lactation in a subject (spontaneously reported to them) that occurs during the trial.

Pregnancies and lactations that occur after the consent form is signed but before treatment allocation/randomization must be reported by the investigator if they cause the subject to be excluded from the trial, or are the result of a protocol-specified intervention, including but not limited to washout or discontinuation of usual therapy, diet, placebo treatment or a procedure.

Pregnancies and lactations that occur from the time of treatment allocation/randomization through 120 days following cessation of Sponsor's product, or 30 days following cessation of treatment if the subject initiates new anticancer therapy, whichever is earlier, must be reported by the investigator. All reported pregnancies must be followed to the completion/termination of the pregnancy. Pregnancy outcomes of spontaneous abortion, missed abortion, benign hydatidiform mole, blighted ovum, fetal death, intrauterine death, miscarriage and stillbirth must be reported as serious events (Important Medical Events). If the pregnancy continues to term, the outcome (health of infant) must also be reported.

Such events must be reported within 24 hours to the Sponsor and within 2 working days to Merck Global Safety. (Attn: Worldwide Product Safety; FAX 215 993-1220)

## 7.2.3 Immediate Reporting of Adverse Events to the Sponsor and to Merck

## 7.2.3.1 Serious Adverse Events

A serious adverse event is any adverse event occurring at any dose or during any use of Merck's product that:

- Results in death;
- Is life threatening;
- Results in persistent or significant disability/incapacity;
- Results in or prolongs an existing inpatient hospitalization;
- Is a congenital anomaly/birth defect;
- Is another important medical event
- <u>Note:</u> In addition to the above criteria, adverse events meeting either of the below criteria, although not serious per ICH definition, are reportable to the Merck in the same timeframe as SAEs to meet certain local requirements. Therefore, these events are considered serious by Merck for collection purposes.
  - Is a new cancer (that is not a condition of the study);

• Is associated with an overdose.

Refer to Table 6.5 for additional details regarding each of the above criteria.

For the time period beginning when the consent form is signed until treatment allocation/randomization, any serious adverse event, or follow up to a serious adverse event, including death due to any cause other than progression of the cancer under study (reference Section 7.2.3.3 for additional details) that occurs to any subject must be reported within 24 hours to the Sponsor and within 2 working days to Merck Global Safety if it causes the subject to be excluded from the trial, or is the result of a protocol-specified intervention, including but not limited to washout or discontinuation of usual therapy, diet, placebo treatment or a procedure.

For the time period beginning at treatment allocation/randomization through 90 days following cessation of treatment, or 30 days following cessation of treatment if the subject initiates new anticancer therapy, whichever is earlier, any serious adverse event, or follow up to a serious adverse event, including death due to any cause other than progression of the cancer under study (reference Section 7.2.3.3 for additional details), whether or not related to the Merck product, must be reported within 24 hours to the Sponsor and within 2 working days to Merck Global Safety.

Additionally, any serious adverse event, considered by an investigator who is a qualified physician to be related to Merck product that is brought to the attention of the investigator at any time following consent through the end of the specified safety follow-up period specified in the paragraph above, or at any time outside of the time period specified in the previous paragraph also must be reported immediately to the Sponsor and to Merck Global Safety.

All subjects with serious adverse events must be followed up for outcome.

# SAE reports and any other relevant safety information are to be forwarded to the Merck Global Safety facsimile number: +1-215-993-1220

A copy of all 15 Day Reports and Annual Progress Reports is submitted as required by FDA, European Union (EU), Pharmaceutical and Medical Devices agency (PMDA) or other local regulators. Investigators will cross reference this submission according to local regulations to the Merck Investigational Compound Number (IND, CSA, etc.) at the time of submission. Additionally investigators will submit a copy of these reports to Merck & Co., Inc. (Attn: Worldwide Product Safety; FAX 215 993-1220) at the time of submission to FDA.

## 7.2.3.2 Events of Clinical Interest

Selected non-serious and serious adverse events are also known as Events of Clinical Interest (ECI) and must be reported within 24 hours to the Sponsor and within 2 working days to Merck Global Safety. (Attn: Worldwide Product Safety; FAX 215 993-1220).

For the time period beginning when the consent form is signed until treatment allocation/randomization, any ECI, or follow up to an ECI, that occurs to any subject must be

reported within 24 hours to the Sponsor and within 2 working days to Merck Global Safety if it causes the subject to be excluded from the trial, or is the result of a protocol-specified intervention, including but not limited to washout or discontinuation of usual therapy, diet, placebo treatment or a procedure.

For the time period beginning at treatment allocation/randomization through 90 days following cessation of treatment, or 30 days following cessation of treatment if the subject initiates new anticancer therapy, whichever is earlier, any ECI, or follow up to an ECI, whether or not related to Merck product, must be reported within 24 hours to the Sponsor and within 24 hours to Merck Global Safety.

Events of clinical interest for this trial include:

- 1. an overdose of Merck product, as defined in Section 7.2.1 Definition of an Overdose for This Protocol and Reporting of Overdose to the Sponsor, that is not associated with clinical symptoms or abnormal laboratory results.
- 2. an elevated AST or ALT lab value that is greater than or equal to 3X the upper limit of normal and an elevated total bilirubin lab value that is greater than or equal to 2X the upper limit of normal and, at the same time, an alkaline phosphatase lab value that is less than 2X the upper limit of normal, as determined by way of protocol-specified laboratory testing or unscheduled laboratory testing.\*

<u>\*Note:</u> These criteria are based upon available regulatory guidance documents. The purpose of the criteria is to specify a threshold of abnormal hepatic tests that may require an additional evaluation for an underlying etiology.

# 7.2.3.3 Protocol-Specific Exceptions to Serious Adverse Event Reporting

Efficacy endpoints as outlined in this section will not be reported to Merck as described in Section 7.2.3- Immediate Reporting of Adverse Events to the Sponsor and to Merck, unless there is evidence suggesting a causal relationship between the drug and the event. Any such event will be submitted to the Sponsor within 24 hours and to Merck Global Safety within 2 working days either by electronic or paper media.

Specifically, the suspected/actual events covered in this exception include any event that is disease progression of the cancer under study.

The Sponsor will monitor unblinded aggregated efficacy endpoint events and safety data to ensure the safety of the subjects in the trial. Any suspected endpoint which upon review is not progression of the cancer under study will be forwarded to Merck Global Safety as a SAE within 2 working days of determination that the event is not progression of the cancer under study

Hospitalization related to convenience (e.g.transportation issues etc.) will not be considered a SAE.

# 7.2.4 Evaluating Adverse Events

An investigator who is a qualified physician will evaluate all adverse events according to the NCI Common Terminology for Adverse Events (CTCAE), version 5.0. Any adverse event which changes CTCAE grade over the course of a given episode will have each change of grade recorded on the adverse event case report forms/worksheets.

All adverse events regardless of CTCAE grade must also be evaluated for seriousness.

Laboratory tests and vital signs which fall out of normal range will only be reported as adverse events if considered clinically significant by the investigator.

Table 6.5 Evaluating Adverse Events

An investigator who is a qualified physician, will evaluate all adverse events as to:

| V4.0 CTCAE<br>Grading | Grade 1 Mild; asymptomatic or mid symptoms; clinical or diagnostic observations only; intervention not indicated. | |
|---|---|---|
| | Grade 2 | Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL. |
| | Grade 3 | Severe or medically significant but not immediately life-threatening; hospitalization or prolongation or hospitalization indicated; disabling; limiting self-care ADL. |
| | Grade 4 | Life threatening consequences; urgent intervention indicated. |
| | Grade 5 | Death related to AE |
| Seriousness | A serious adv | verse event is any adverse event occurring at any dose or during any use of Merck product that: |
| | †Results in d | leath; or |
| | †Is life threatening; or places the subject, in the view of the investigator, at immediate risk of death from the event as it occurred (Note: This does not include an adverse event that, had it occurred in a more severe form, might have caused death.); or | |
| | †Results in a | persistent or significant disability/incapacity (substantial disruption of one's ability to conduct normal life functions); or |
| | hospitalizatio<br>worsened is r | or prolongs an existing inpatient hospitalization (hospitalization is defined as an inpatient admission, regardless of length of stay, even if the on is a precautionary measure for continued observation. (Note: Hospitalization for an elective procedure to treat a pre-existing condition that has not not a serious adverse event. A pre-existing condition is a clinical condition that is diagnosed prior to the use of a Merck product and is documented in medical history.); or |
| | †Is a congen | ital anomaly/birth defect (in offspring of subject taking the product regardless of time to diagnosis);or |
| | Is a new cancer (that is not a condition of the study) (although not serious per ICH definition, is reportable to the Sponsor within 24 hours and to Merck within 2 working days to meet certain local requirements); or | |
| | <b>Is an overdose</b> (whether accidental or intentional). Any adverse event associated with an overdose is considered a serious adverse event for collection purposes. An overdose that is not associated with an adverse event is considered a non-serious event of clinical interest and must be reported within 24 hours to the Sponsor and to Merck within 2 working days | |
| | | rtant medical events that may not result in death, not be life threatening, or not require hospitalization may be considered a serious adverse event when, appropriate medical judgment, the event may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes |

| | listed previously (designated above by a †). | |
|---|---|---|
| Duration | Record the start and stop dates of the adverse event. If less than 1 day, indicate the appropriate length of time and units | |
| Action taken | Did the adverse event cause Merck product to be discontinued? | |
| Relationship to<br>Merck Product | | |
| | Exposure Time Course | Is there evidence that the subject was actually exposed to Merck product such as: reliable history, acceptable compliance assessment (pill count, diary, etc.), expected pharmacologic effect, or measurement of drug/metabolite in bodily specimen? Did the AE follow in a reasonable temporal sequence from administration of Merck product? Is the time of onset of the AE compatible with a drug-induced effect (applies to trials with investigational medicinal product)? |
| | Likely Cause | Is the AE not reasonably explained by another etiology such as underlying disease, other drug(s)/vaccine(s), or other host or environmental factors |

| Relationship | The following | The following components are to be used to assess the relationship between the test drug and the AE: (continued) |
|---|---|---|
| to Merck<br>Product | Dechallenge Was Merck product discontinued or dose/exposure/frequency reduced? | |
| (continued) | | If yes, did the AE resolve or improve? |
| (continued) | | If yes, this is a positive dechallenge. If no, this is a negative dechallenge. |
| | | (Note: This criterion is not applicable if: (1) the AE resulted in death or permanent disability; (2) the AE resolved/improved despite continuation of the Sponsor's product; or (3) the trial is a single-dose drug trial); or (4) Sponsor's product(s) is/are only used one time.) |
| | Rechallenge | Was the subject re-exposed to Merck product in this study? |
| | | If yes, did the AE recur or worsen? |
| | | If yes, this is a positive rechallenge. If no, this is a negative rechallenge. |
| | | (Note: This criterion is not applicable if: (1) the initial AE resulted in death or permanent disability, or (2) the trial is a single-dose drug trial); or (3) Sponsor's product(s) is/are used only one time). |
| | | NOTE: IF A RECHALLENGE IS PLANNED FOR AN ADVERSE EVENT WHICH WAS SERIOUS AND WHICH MAY HAVE BEEN CAUSED BY MERCK PRODUCT, OR IF REEXPOSURE TO MERCK PRODUCT POSES ADDITIONAL POTENTIAL SIGNIFICANT RISK TO THE SUBJECT, THEN THE RECHALLENGE MUST BE APPROVED IN ADVANCE BY THE SPONSOR AS PER DOSE MODIFICATION GUIDELINES IN THE PROTOCOL. |
| | Consistency<br>with Trial<br>Treatment<br>Profile | Is the clinical/pathological presentation of the AE consistent with previous knowledge regarding Merck product or drug class pharmacology or toxicology? |
| | of relationship will<br>the above elements | be reported on the case report forms /worksheets by an investigator who is a qualified physician according to his/her best clinical judgment, including s. |
| Record one of the following | | Use the following scale of criteria as guidance (not all criteria must be present to be indicative of Merck product relationship). |
| Yes, there is a reasonable possibility of Merck product relationship. | | There is evidence of exposure to Merck product. The temporal sequence of the AE onset relative to the administration of Merck product is reasonable. The AE is more likely explained by Merck product than by another cause. |
| | | Subject did not receive the Merck product OR temporal sequence of the AE onset relative to administration of Merck product is not reasonable OR the AE is more likely explained by another cause than the Merck product. (Also entered for a subject with overdose without an associated AE.) |

## 7.2.5 Sponsor Responsibility for Reporting Adverse Events

All Adverse Events will be reported to regulatory authorities, IRB/IECs and investigators in accordance with all applicable global laws and regulations.

## 8.0 STATISTICAL ANALYSIS PLAN

## 8.1 Statistical Analysis Plan Summary

Simon two-stage single-arm phase II study

## 8.2 Statistical Analysis Plan

This will be a standard phase II study. The sample size calculation is based on the assumption that a true response of >38% would generate interest in a larger randomized study. With 35 patients we will be able to test the hypothesis that the true response rate is 38% versus 18% (null) with a power of 90% and a type 1 error of 8%. Patients will be accrued to the protocol according to a Simon's two-stage minimax design. 20 patients will be enrolled in stage 1. If 4 or more responses are observed, than another 15 subjects will be enrolled into stage 2. At the completion of the study, if 10 or more responses out of N=35 are observed, significance at 8% is reached. Under this design, if the true response rate is  $\geq 38\%$ , then the probability of observing  $\geq 1$  response in stage 1 is 95%.

The progression-free survival (PFS) estimates will be shown by Kaplan-Meier curve, and noted at landmark times: 3, 6, and 12 months. For patients with a response, the duration of response will be plotted using a Kaplan-Meier curve and the median survival obtained from it. The progression-free survival estimates will be shown by Kaplan-Meier curve, and noted at landmark times: 3, 6, and 12 months. The overall survival (OS) estimates will be shown by Kaplan-Meier curve, and noted at landmark times, such as: median and 12 months. Overall safety will be assessed by identifying the highest toxicity grade for each patient; this will also be done for selected key toxicities.

# 9.0 LABELING, PACKAGING, STORAGE AND RETURN OF CLINICAL SUPPLIES

## 9.1 Investigational Product

The investigator shall take responsibility for and shall take all steps to maintain appropriate records and ensure appropriate supply, storage, handling, distribution and usage of investigational product in accordance with the protocol and any applicable laws and regulations.

Clinical Supplies will be provided by Merck as summarized in Table 7.

Table 7 Product Descriptions

| Product Name & Potency | Dosage Form |
|---------------------------|----------------------------------|
| Pembrolizumab 50 mg | Lyophilized Powder for Injection |
| Pembrolizumab 100 mg/ 4mL | Solution for Injection |
| Lenvatinib 10 mg | Hard hypromellose capsules |
| Lenvatinib 4mg | Hard hypromellose capsules |

# 9.2 Packaging and Labeling Information

Clinical supplies will be affixed with a clinical label in accordance with regulatory requirements.

# 9.3 Clinical Supplies Disclosure

This trial is open-label; therefore, the subject, the trial site personnel, the Sponsor and/or designee are not blinded to treatment. Drug identity (name, strength) is included in the label text; random code/disclosure envelopes or lists are not provided.

# 9.4 Storage and Handling Requirements

Clinical supplies must be stored in a secure, limited-access location under the storage conditions specified on the label.

Receipt and dispensing of trial medication must be recorded by an authorized person at the trial site.

Clinical supplies may not be used for any purpose other than that stated in the protocol.

## 9.5 Returns and Reconciliation

The investigator is responsible for keeping accurate records of the clinical supplies received from Merck or designee, the amount dispensed to and returned by the subjects and the amount remaining at the conclusion of the trial.

Upon completion or termination of the study, all unused and/or partially used investigational product will be destroyed at the site per institutional policy. It is the Investigator's responsibility to arrange for disposal of all empty containers, provided that procedures for proper disposal have been established according to applicable federal, state, local and institutional guidelines and procedures, and provided that appropriate records of disposal are kept.

## 10.0 ADMINISTRATIVE AND REGULATORY DETAILS

# 10.1 Compliance with Trial Registration and Results Posting Requirements

Under the terms of the Food and Drug Administration Modernization Act (FDAMA) and the Food and Drug Administration Amendments Act (FDAAA), the Sponsor of the trial is solely responsible for determining whether the trial and its results are subject to the requirements for submission to the Clinical Trials Data Bank, http://www.clinicaltrials.gov. Information posted will allow subjects to identify potentially appropriate trials for their disease conditions and pursue participation by calling a central contact number for further information on appropriate trial locations and trial site contact information.

# 10.2 Data Management

The investigator must prepare and maintain adequate and accurate case histories designed to record all observations and other data pertinent to the study for each research participant. This information enables the study to be fully documented and the study data to be subsequently verified.

Original source documents supporting entries in the case report forms include but are not limited to hospital records, clinical charts, laboratory and pharmacy records, recorded data from automated instruments, microfiches, photographic negatives, microfilm or magnetic media, and/or x-rays.

The trial will be monitored per Moffitt Cancer Center policy MRI-P.PSO.03, *Monitoring of Investigator Initiated Clinical Research*. Data will be captured in Oncore, Moffitt's Clinical Trials Database, Regulatory documents and case report forms will be monitored internally according to Moffitt Cancer Center Monitoring Policies. Monitoring will be performed regularly to verify data is accurate, complete and verifiable from source documents; and the conduct of the trial is in compliance with the currently approved protocol/amendments, Good Clinical Practice, and applicable regulatory requirements

Retained records will include all documentation of adverse events, records of study drug receipt and dispensation, and all IRB correspondence for at least 5 years after the investigation is completed.

### 11.0 APPENDICES

### 11.1 ECOG Performance Status

| Grade | Description |
|---|---|
| 0 | Normal activity. Fully active, able to carry on all pre-disease |
| U U | performance without restriction. |
| | Symptoms, but ambulatory. Restricted in physically strenuous |
| 1 | activity, but ambulatory and able to carry out work of a light or |
| | sedentary nature (e.g., light housework, office work). |
| | In bed <50% of the time. Ambulatory and capable of all self-care, |
| 2 | but unable to carry out any work activities. Up and about more than |
| | 50% of waking hours. |
| 3 | In bed >50% of the time. Capable of only limited self-care, confined |
| 3 | to bed or chair more than 50% of waking hours. |
| 4 | 100% bedridden. Completely disabled. Cannot carry on any self- |
| | care. Totally confined to bed or chair. |
| 5 | Dead. |

<sup>\*</sup>As published in Am. J. Clin. Oncol.: Oken, M.M., Creech, R.H., Tormey, D.C., Horton, J., Davis, T.E., McFadden, E.T., Carbone, P.P.: Toxicity And Response Criteria Of The Eastern Cooperative Oncology Group. Am J Clin Oncol 5:649-655, 1982. The Eastern Cooperative Oncology Group, Robert Comis M.D., Group Chair.

## 11.2 Common Terminology Criteria for Adverse Events V4.0 (CTCAE)

The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for adverse event reporting. (http://ctep.cancer.gov/reporting/ctc.html)

# 11.3 Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 Criteria for Evaluating Response in Solid Tumors

RECIST version 1.1\* will be used in this study for assessment of tumor response. While either CT or MRI may be utilized, as per RECIST 1.1, CT is the preferred imaging technique in this study.

E.A. Eisenhauer, P. Therasse, J. Bogaerts, L.H. Schwartz, D. Sargent, R. Ford, J. Dancey, S. Arbuck, S. Gwyther, M. Mooney, L. Rubinstein, L. Shankar, L. Dodd, R. Kaplan, D. Lacombe, J. Verweij. New response evaluation criteria in solid tumors: Revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47.

<sup>\*</sup> As published in the European Journal of Cancer:

#### 12.0 REFERENCES

- 1. LENVIMA (lenvatinib) Package Insert. In: FDA, ed. FDA 2015.
- 2. Strosberg J, El-Haddad G, Wolin E, et al. Phase 3 Trial of (177)Lu-Dotatate for Midgut Neuroendocrine Tumors. N Engl J Med 2017;**376**(2):125-35 doi: 10.1056/NEJMoa1607427[published Online First: Epub Date]|.
- 3. Caplin ME, Pavel M, Cwikla JB, et al. Lanreotide in metastatic enteropancreatic neuroendocrine tumors. N Engl J Med 2014;**371**(3):224-33 doi: 10.1056/NEJMoa1316158[published Online First: Epub Date]|.
- 4. Pavel ME, Baudin E, Oberg KE, et al. Efficacy of everolimus plus octreotide LAR in patients with advanced neuroendocrine tumor and carcinoid syndrome: final overall survival from the randomized, placebo-controlled phase 3 RADIANT-2 study. Ann Oncol 2017;28(7):1569-75 doi: 10.1093/annonc/mdx193[published Online First: Epub Date]|.
- 5. Yao JC, Fazio N, Singh S, et al. Everolimus for the treatment of advanced, non-functional neuroendocrine tumours of the lung or gastrointestinal tract (RADIANT-4): a randomised, placebo-controlled, phase 3 study. Lancet 2016;**387**(10022):968-77 doi: 10.1016/S0140-6736(15)00817-X[published Online First: Epub Date]].
- 6. Raymond E, Dahan L, Raoul JL, et al. Sunitinib malate for the treatment of pancreatic neuroendocrine tumors. N Engl J Med;**364**(6):501-13 doi: 10.1056/NEJMoa1003825[published Online First: Epub Date]|.
- 7. Strosberg JR, Fine RL, Choi J, et al. First-line chemotherapy with capecitabine and temozolomide in patients with metastatic pancreatic endocrine carcinomas. Cancer 2011;117(2):268-75 doi: 10.1002/cncr.25425[published Online First: Epub Date]|.
- 8. Capdevila Castillon J, Fazio N, Lopez C, et al. Efficacy of Lenvatinib in patients with advanced pancreatic (panNETs) and gastrointestinal (giNETs) grade 1/2 (G1/G2) neuroendocrine tumors. ESMO 2018. Munich, Germany, 2018.
- 9. Amin A, Plimack ER, Ernstoff MS, et al. Safety and efficacy of nivolumab in combination with sunitinib or pazopanib in advanced or metastatic renal cell carcinoma: the CheckMate 016 study. J Immunother Cancer 2018;6(1):109 doi: 10.1186/s40425-018-0420-0[published Online First: Epub Date]|.
- 10. Choueiri TK, Larkin J, Oya M, et al. Preliminary results for avelumab plus axitinib as first-line therapy in patients with advanced clear-cell renal-cell carcinoma (JAVELIN Renal 100): an open-label, dose-finding and dose-expansion, phase 1b trial. Lancet Oncol 2018;19(4):451-60 doi: 10.1016/S1470-2045(18)30107-4[published Online First: Epub Date]|.
- 11. McDermott DF, Huseni MA, Atkins MB, et al. Clinical activity and molecular correlates of response to atezolizumab alone or in combination with bevacizumab versus sunitinib in renal cell carcinoma. Nat Med 2018;**24**(6):749-57 doi: 10.1038/s41591-018-0053-3[published Online First: Epub Date]|.
- 12. Iyer PC, Dadu R, Gule-Monroe M, et al. Salvage pembrolizumab added to kinase inhibitor therapy for the treatment of anaplastic thyroid carcinoma. J Immunother Cancer 2018;6(1):68 doi: 10.1186/s40425-018-0378-y[published Online First: Epub Date]|.